CLINICAL TRIAL: NCT03360565
Title: Obesity: Prospective Evaluation of Upper Airway Obstruction and Compliance in Obese Patients in Pre and Post Bariatric Surgery : A Monocentric Observational Study
Brief Title: Obesity: Prospective Evaluation of Upper Airway Obstruction and Compliance in Obese Patients in Pre and Post Bariatric Surgery
Acronym: OBANEZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A02883-50
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Obstructive Sleep Apnea Syndrome (OSAS)
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This clinical trial is a monocentric, prospective, observational and controlled trial (historical cohort control group of healthy non-obese subjects who had Nasal functional exploration for Snoring) as part of current care.

This study concerns the prevalence of obstructive sleep apnea syndrome (OSAS). OSAS is elevated in subjects with morbid obesity (BMI≥40) (on average 70%). International recommendations agree on the need to seek OSAS before bariatric surgery because of the high risk of complications.

Increased nasal resistance could also be related to a limitation of inspiratory flow due to an abnormality of the elasticity of the nasal mucosa or "nasal compliance". Adipose infiltration of the nasal mucosa may occur during obesity.

These tissue changes (decreased vaso-erectile tissue and increased adipose tissue) could modify the nasal compliance, which the decrease would be a possible factor of severity of OSAS in obese patients. Screening for an abnormality of compliance could also anticipate a difficulty of equipment for Continuous Positive Airway Pressure (CPAP) in the case of associated OSAS.

All patients who must have bariatric surgery and get in the criteria are included. They will have to do a medical checkup pre and post-operative (polygraphy + ear/nose/throat assessment (ENT) + Nasal functional exploration). They will be followed for 13 to 24 months.

The main objective of this research is to demonstrate a reduction of at least 30% of nasal compliance in a group of obese subjects (BMI> 35) compared to a control group of healthy subjects.

The secondary objectives are to is to demonstrate an increase of 30% in resistance in patients with BMI> 35 compared to control group and a normalization of nasal compliance 1 year after surgery when their weight is normalized (BMI <30).

A study period of 4 years is planned.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary Patient
* Patients aged 18 years or older.
* BMI > 35
* Patient included in the bariatric surgery protocol
* Medical checkup :polygraphy and Respiratory Functional Exploration (RFE)

Exclusion Criteria:

* Impossible to obtain a consent or age less than 18 years
* Heart / Kidney Failure
* Absence of affiliation to a Social Security scheme
* History of rhinological surgery
* Pregnancy, Breastfeeding
* Subject presenting a congenital or acquired obstructive nasal obstructive physical obstacle (obstructive deviation, craniofacial malformation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participation to the study will be proposed to all patients who must have bariatric surgery and have a preoperative assessment
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-03-02 (Actual); Primary Completion 2018-03-02 (Estimated); Study Completion 2020-03-02 (Estimated)

PRIMARY OUTCOMES:
To demonstrate a reduction of at least 30% of nasal compliance in a group of obese subjects (BMI> 35) compared to a control group of healthy subjects | before bariatric surgery

SECONDARY OUTCOMES:
To demonstrate an increase of 30% in resistance in patients with BMI> 35 compared to control group | before bariatric surgery
To demonstrate a normalization of nasal compliance when the weight is normalized (BMI <30) | 9 month (+3month) after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emilie BEQUIGNON, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France